CLINICAL TRIAL: NCT04853134
Title: Proxalutamide Treatment for COVID-19 Female Outpatients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was combined with another study
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-DRUG-SARS-005
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-04

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: Proxalutamide; Androgens
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — proxalutamide; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Placebo Comparator): Standard of care as determined by the PI
  Interventions: Other: Standard of Care
- Proxalutamide + Standard Care (Active Comparator): Proxalutamide + standard of care as determined by the PI
  Interventions: Drug: Proxalutamide

INTERVENTIONS:
Drug: Proxalutamide — 200 mg q.d.
  Arms: Proxalutamide + Standard Care
Other: Standard of Care — Standard of care as determined by the PI
  Arms: Standard Care

SUMMARY:
This study is intended to explore the possible protective role of anti-androgens in SARS-CoV-2 infection

DETAILED DESCRIPTION:
During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%).Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2). TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro. Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene. In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor. Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males.

Androgenetic alopecia (AGA), often referred to as male pattern hair loss, is the most common form of hair loss among men. The development of androgenetic alopecia is androgen mediated and is dependent on genetic variants found in the androgen receptor gene located on the X chromosome; thus, it is hypothesized that men with AGA would be more prone to severe COVID-19 disease. The investigators conducted a preliminary observational study of hospitalized COVID-19 patients at two Spanish tertiary hospitals between March 23-April 6, 2020 to test this theory. In total, 41 Caucasian males admitted to the hospitals with a diagnosis of bilateral SARS-CoV-2 pneumonia were analyzed. The mean age of patients was 58 years (range 23-79). Among them, 29 (71%) were diagnosed with AGA (16 (39%) were classified as severe AGA (Hamilton IV or above)) and 12 (29%) did not present clinical signs of AGA. The diagnosis of AGA was performed clinically by a dermatologist. The precise prevalence of AGA among otherwise healthy Spanish Caucasian males is unknown; however, based on published literature, the expected prevalence of a similar age-matched Caucasian population is approximately 31-53%.

Based on the scientific rationale combined with this preliminary observation, the investigators propose to test an anti-androgen as a treatment for patients recently diagnosed with COVID-19.

We have chosen the use of the novel second generation androgen receptor (AR) antagonist proxalutamide as a means for rapid reduction in AR activity. Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells.

This study is intended to explore the possible protective role of anti-androgens in SARS-CoV-2 infection. Provided anti-androgens are effective in reducing the rate of COVID-19 hospitalization, subjects enrolled in this study may experience a lower rate of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Female age >=18 years old
* Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization
* Clinical status on the NIAID COVID-19 Ordinal Scale of 1 or 2 (i.e., not requiring hospitalization)
* Coagulation: INR<=1.5XULN, and APTT<=1.5XULN
* Subject (or legally authorized representative) gives written informed consent prior to any study screening procedures
* Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study
* Not Pregnant or breastfeeding

Exclusion Criteria:

* Subject enrolled in a study to investigate a treatment for COVID-19 Page 17 of 40
* Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc...
* Patients who are allergic to the investigational product or similar drugs (or any excipients)
* Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
* Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
* Subjects with uncontrolled medical conditions that could compromise participation in the study (e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
* Known diagnosis of human immunodeficiency virus (HIV) , hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory)
* Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
* Estimated glomerular filtration rate (eGFR) < 30 ml/min
* Severe kidney disease requiring dialysis
* Subject unlikely to return for day 15 site visit for reasons other then remission
* Subject (or legally authorized representative) not willing or unable to provide informed consent
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a study in female subjects as an extension to NCT04446429 for male subjects
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 hospitalization | 30 days
  Percentage of subjects hospitalized due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Cadegiani, MD, Principal Investigator — Corpometria Institute; Carlos Wambier, MD, Principal Investigator — Applied Biology, Inc.; Andy Goren, MD, Study Director — Applied Biology, Inc.
Locations (1):
- Corpometria Institute, Brasília, Brazil